CLINICAL TRIAL: NCT04811794
Title: Young Survivors at Kantonsspital Aarau, Switzerland - A Standardized Assessment of Long-Term and Late-Onset Health Events in Survivors of Childhood and Adolescent Cancer
Brief Title: Young Survivors at Kantonsspital Aarau, Switzerland
Status: Recruiting | Type: Observational
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Katrin Scheinemann, Division Head of Pediatric Oncology-Hematology, Kantonsspital Aarau
Other Study IDs: AO_2020-00012
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Childhood Cancer; Late Effects
Keywords: Childhood Cancer; Survivor; Late Effects; CTCAE
MeSH Terms: conditions — Neoplasms | interventions — Restraint, Physical; Health Records, Personal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (largest part of the cohort): Children, adolescents, and adults who are still in follow-up care (data are collected retrospectively until 2016 at the most)
  Interventions: Other: Physical examination, diagnostic tests, laboratory tests; Other: Personal history
- Group B (very small part of the cohort): Children, adolescents, and adults who left follow-up care (data are collected retrospectively until 2016 at the most)
  Interventions: Other: Physical examination, diagnostic tests, laboratory tests; Other: Personal history

INTERVENTIONS:
Other: Physical examination, diagnostic tests, laboratory tests — Physical examination, diagnostic tests (e.g. lung function test, echocardiography, audiometry), and laboratory tests (e.g. kidney parameter, hormonal levels) depend on examined organ system.
Other: Personal history — Personal history on diagnosis, treatment, and socioeconomic factors

SUMMARY:
The Young Survivors at Kantonsspital Aarau project assesses the prevalence and severity of late effects in survivors of childhood and adolescent cancer according to the modified CTCAE criteria prospectively. The clinical data are generated during regular follow-up care visits, the collection starts directly after completion of treatment and is longitudinally.

DETAILED DESCRIPTION:
Background:

Around 250-300 children and adolescents below the age of 21 years are newly diagnosed with cancer in Switzerland every year. Research led to remarkable progress in survival in the last decades. The 10-year survival rate in Switzerland is currently 87%. Previous research showed that, depending on the treatment exposure, a high proportion of these survivors suffer from chronic medical conditions, so called late effects.

Many studies on late effects in former childhood cancer patients are based on retrospective data. However, this type of study design has unavoidable limitations, such as missing data, different coding and grading of severity of late effects, and the assessment at different time points. Therefore, we need prospectively collected data, including severity coding in a standardized way, to overcome these limitations.

Objectives:

The overarching aim of "Young Survivors at Kantonsspital Aarau, Switzerland" is to assess late effects in childhood cancer survivors prospectively and in a standardized way. These data will contribute to the increasing knowledge on long-term outcomes and late effects in the future. This new knowledge is important in order to be able to adapt and improve long-term follow-up care. In the longer term, survivors will benefit from this extensive and prospective data collection.

Methods:

"Young Survivors at Kantonsspital Aarau" has a registry-like design. Data produced during regular follow-up visits are collected in a comprehensive database and in a standardized way. We collect all information generated prospectively from start of the study onwards and retrospectively until January 2016. From 2016 onward, all medical records are kept electronically. We classify and grade the severity of late effects according to the modified National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.03). The outcome variables correspond to results from risk-stratified organ examinations, which are performed according to the Children's Oncology Group guidelines v5.0. The exposure variables correspond to information from the patients' medical history, including detailed information on cancer diagnosis and treatment. The data will be analyzed in an exposure- or organ system-driven approach. We start recruitment with patients diagnosed and treated at the Kantonsspital Aarau. The design of the study allows the inclusion of other clinics in the future.

Research and significance:

Research on late effects of former childhood cancer patients often relies on retrospective data collection, which is associated with unpreventable limitations. "Young Survivors at Kantonsspital Aarau" overcomes these limitations and additionally grades the severity of late effects in a standardized way. This allows us to analyze changes in severity of late effects over time, within and between survivors. This information will increase our knowledge on late effects and contribute to long-term follow-up care.

ELIGIBILITY:
Inclusion Criteria:

Group A:

Children and adolescents who:

* have been treated for cancer in the Division of Oncology-Hematology, Department of Pediatrics, at the Kantonsspital Aarau,
* have been diagnosed at age 0-18 years,
* are still in regular follow-up care at the Kantonsspital Aarau,
* have finished cancer treatment and entered follow-up care, and
* signed informed consent

Group B:

Adolescents and adults who:

* fulfill the same inclusion criteria as Group A
* are not in regular follow-up care anymore

Exclusion Criteria:

Childhood Cancer Survivors who:

* are in a palliative situation or
* have not given consent for further use of medical data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes all children, adolescents and adults who have been treated for cancer in the Division of Oncology-Hematology, Department of Pediatrics, at the Kantonsspital Aarau and who have completed their treatment and have entered follow-up care.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2071-03-15 (Estimated); Study Completion 2072-03-15 (Estimated)

PRIMARY OUTCOMES:
Test results to assess organ-specific late effects (example of cardiac health) | at recruitment or 2016 onwards, whichever comes first
  Number of survivors with heart valve disorder, hypertension, left ventricular systolic dysfunction when at risk for cardiac late effects

SECONDARY OUTCOMES:
Test results to assess organ-specific late effects (example of cardiac health) | annually from recruitment or 2016 onwards, whichever comes first
  Number of survivors with heart valve disorder, hypertension, left ventricular systolic dysfunction etc. when at risk for cardiac late effects
Sociodemographic and socioeconomic characteristics (e.g. age at clinical examination, gender, education or working situation, living situation) | annually from recruitment or 2016 onwards, whichever comes first
Comorbidities (e.g. arterial hypertension, obesity) as risk factors for late effects | annually from recruitment or 2016 onwards, whichever comes first
Diagnosis-related data (e.g. age at diagnosis, diagnosis, disease stage, treatment protocol) | at recruitment or 2016 onwards, whichever comes first
Treatment-related data (e.g. cumulative doses of chemotherapy and radiotherapy, surgery, hematopoietic stem cell transplantation ) | at recruitment or 2016 onwards, whichever comes first

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Oncology - Hematology, Department of Pediatrics, Kantonsspital Aarau, Aarau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Otth M, Drozdov D, Hugli C, Scheinemann K. Young Survivors at KSA: registry for standardised assessment of long-term and late-onset health events in survivors of childhood and adolescent cancer-a study protocol. BMJ Open. 2021 Dec 3;11(12):e053749. doi: 10.1136/bmjopen-2021-053749. PMID 34862296